CLINICAL TRIAL: NCT04487821
Title: EFFECTS OF VESTIBULAR REHABILITATION THERAPY (VRT) ON BALANCE, SPEED AND AGILITY IN POST-CONCUSSION FOOTBALL PLAYERS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zohra Institute of Health Sciences (Other)
Responsible Party: Principal Investigator, Syed Alamdar Hussain, Syed Alamdar Hussain, Zohra Institute of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZIHS-1205/MS/12
Record Dates: First submitted 2020-07-23; First posted 2020-07-27 (Actual); Last update posted 2020-07-27 (Actual); Status verified 2020-07

CONDITIONS: Concussion, Mild
Keywords: Traumatic Brain Injury; Concussion; Vestibular Rehabilitation Therapy; Football; Balance
MeSH Terms: conditions — Brain Concussion; Brain Injuries, Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Subjects were randomly assigned and informed consent was obtained, the subjects were educated about treatment. This contained 4 types of progressive activities. Respectively every type contains 2 to 4 tasks, performed in sets of 10 repetitions for 4 weeks.
  Results were obtained by using Balance scoring system, and physical performance test for speed and agility
  Interventions: Other: Cawthorne Cooksey Exercises
- Control Group (No Intervention): Control group: (Group B) Subjects were randomly assigned and informed consent was obtained, the subjects were educated about treatment. They were asked to perform the regular drills.
  Results were obtained using Balance Error scoring system and physical performance test for speed and agility.

INTERVENTIONS:
Other: Cawthorne Cooksey Exercises — Activity sitting on the "Exercise Ball" swing (eye movements, first slow and then fast)
  Swing sitting activity (head movements, first slow then fast - eyes open and eyes closed)
  Trunk activities focusing on balance
  Dynamic balance activity focusing on standing
  Arms: Experimental Group

SUMMARY:
Traumatic brain injury (TBI) is one and utmost rampant attained neurological conditions which can happen in young adults. Vestibular Rehabilitation Therapy can help them improve their balance, speed and agility.

DETAILED DESCRIPTION:
Total 40 sample size out of which were divided into control and experimental group. Concussed football athletes with age ranging 15-25 year, those participating actively in the sports were included in the study in the region of Kyber Pukhtoonkhwa Peshawar.

ELIGIBILITY:
Inclusion Criteria:

Active Male football player. Age between 15-25 years. Known cases of concussion were included in the study. Those patients complaining mild vertigo & participating in sports

Exclusion Criteria:

Concussion other than sports. History of metabolic diseases. History of recent fractures.

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Balance | upto 8 weeks
  Balance Error Scoring System (BESS) which us used to evaluate the balance of the athlete
Agility | upto 8 weeks
  30 Ft Agility Shuttle Run which is used to evaluate agility of athletes
Speed | upto 8 weeks
  30 Meter dash which is used to evaluate the speed of the athlete

CONTACTS AND LOCATIONS:
Locations (1):
- Syed Alamdar Hussain, Peshawar, Khyber Pakhtunkhwa, Pakistan